CLINICAL TRIAL: NCT07348003
Title: Examining the Effectiveness of Single-Limb Exercise Training for COPD Patients During Exacerbation Periods
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alper Kemal Gürbüz (Other)
Responsible Party: Sponsor-Investigator, Alper Kemal Gürbüz, research assistant, Kırıkkale University
Organization: Kırıkkale University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GurbuzTez
Record Dates: First submitted 2025-12-29; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Chronic Obstructive Airways Disease Exacerbated
Keywords: copd; exacerbated; exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study is an interventional clinical trial designed to evaluate the effects of an exercise therapy program. Participants will be prospectively assigned to one of two study arms: an intervention group and a control group.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Active Comparator): Single-Limb Resistance Exercise Group: Participants will perform unilateral resistance exercises for six major muscle groups (shoulder flex/abd, elbow flex, hip flex, knee flex/ext) using free weights in a seated position.
  Interventions: Other: Single Limb Exercise Training; Other: Routine Exercise
- Control Group (Other): Routine Physiotherapy Intervention: The control group will undergo standard inpatient physiotherapy, including breathing retraining (diaphragmatic and pursed-lip breathing) and thoracic expansion exercises.
  Interventions: Other: Routine Exercise

INTERVENTIONS:
Other: Single Limb Exercise Training — Participants will perform unilateral resistance exercises for six major muscle groups (shoulder flex/abd, elbow flex, hip flex, knee flex/ext) using free weights in a seated position. The intensity is set at 50-70% of 1RM, consisting of 2 sets of 8 repetitions per limb. This 8-week program will be conducted twice weekly as an adjunct to routine hospital physiotherapy and standard inpatient physiotherapy, including breathing retraining (diaphragmatic and pursed-lip breathing) and thoracic expansion exercises.
  Arms: Exercise group
Other: Routine Exercise — Physiotherapy Intervention: Just standard inpatient physiotherapy, including breathing retraining (diaphragmatic and pursed-lip breathing) and thoracic expansion exercises.

SUMMARY:
Resistance exercise applications during acute exacerbations of Chronic Obstructive Pulmonary Disease (COPD) are employed to enhance functional capacity and prevent muscle atrophy by increasing muscle strength.

Owing to the limited cardiorespiratory reserve of COPD patients, single-limb exercises are better tolerated compared to traditional bilateral exercises. A study conducted by Vogiatzis et al. (2009) indicated that single-leg exercises require lower ventilation and result in more efficient oxygen consumption than bilateral exercises. This physiological advantage may be effective in reducing muscle weakness by increasing exercise endurance in COPD patients with restricted respiratory capacity.

The present study aims to demonstrate that single-limb resistance exercise is an effective rehabilitation method for increasing functional exercise capacity in patients during COPD exacerbations compared to a control group. Furthermore, the therapeutic effects of single-limb resistance exercises on dyspnea perception, fatigue, anxiety, and depression will be established. The study will also show that these exercises are both feasible and safe within rehabilitation protocols during the exacerbation period.

DETAILED DESCRIPTION:
Pathophysiology and Rehabilitation in Acute Exacerbation of COPD An acute exacerbation of Chronic Obstructive Pulmonary Disease (COPD) represents an acute process that accelerates disease progression and exerts systemic effects. This period is characterized by a sudden worsening of primary symptoms, such as dyspnea, increased sputum volume, and heightened sputum viscosity. Exacerbations lead to increased hospitalization rates, diminished quality of life, and elevated mortality among COPD patients. According to the GOLD 2024 report, a COPD exacerbation is defined as an event characterized by increased dyspnea, cough, and sputum that develops in less than 14 days and necessitates a change in treatment. These episodes are generally attributed to increased airway infection, environmental pollution, or other inflammatory triggers.

During these periods, respiratory functions decline acutely, leading to impaired oxygenation and physiological stress. Research indicates a significant decrease in skeletal muscle function during exacerbations, with muscle weakness becoming a prominent clinical feature. This acute weakness develops due to various factors, including systemic inflammation, nutritional deficiencies, and the use of corticosteroids. Observations show a reduction in myoblast determination proteins and insulin-like growth factor-I levels in skeletal muscle during the exacerbation process; this suggests that physical inactivity is a critical factor in acute muscle dysfunction.

Most patients face conditions requiring inactivity, such as bed rest, during an exacerbation. Inactivity causes a rapid decline in muscle strength, particularly in older individuals; one study demonstrated that 10 days of bed rest resulted in a 15% reduction in quadriceps strength. Under stressful conditions, this effect becomes even more pronounced, and medications such as corticosteroids can exacerbate the detrimental effects of inactivity. Limitation of physical activity during this period both accelerates skeletal muscle loss and adversely affects the long-term mobilization capabilities of patients.

Treatment during a COPD exacerbation aims to alleviate symptoms and improve quality of life. Management typically involves bronchodilators (β2-agonists and anticholinergics), inhaled corticosteroids, and antibiotics. Furthermore, systemic corticosteroids can rapidly improve symptoms by suppressing inflammation. Approaches such as pulmonary rehabilitation, exercise, and breathing techniques can reduce dyspnea by increasing functional capacity . Non-invasive positive pressure ventilation (NIPPV) is utilized for patients experiencing severe respiratory distress. To prevent infections, influenza and pneumococcal vaccinations are recommended, while smoking cessation and avoiding air pollution also reduce the risk of exacerbation.

Exercise performed during a COPD exacerbation helps patients maintain physical capacity and accelerates the recovery process. However, exercises during this period must be meticulously planned, as acute exacerbations lead to impaired respiratory function and increased systemic inflammation. Exercise interventions are typically initiated at low intensity to preserve cardiorespiratory function, support muscle strength, and ensure general mobility.

Low-intensity cardiorespiratory endurance exercises, such as walking or stationary cycling, are recommended during the exacerbation period. These exercises improve oxygenation in skeletal muscles. A study by Vaes et al. (2017) stated that low-intensity cardio exercises initiated during a COPD exacerbation are effective in preserving functional capacity. During an exacerbation, weakness may be observed particularly in the lower extremities, such as the quadriceps. Lower extremity exercises initiated at low resistance levels help patients maintain muscle function and reduce skeletal muscle loss. The study by Greening et al. showed that low-intensity resistance exercises during the exacerbation period are safe and effective for increasing muscle strength .

In COPD, single-limb exercises are implemented to increase tolerance to physical activity and preserve muscle strength, especially during the exacerbation period. These exercises aim to work muscle groups in isolation by focusing on one limb, thereby minimizing energy consumption and reducing the risk of exercise intolerance. During single-limb exercises, muscles operate with lower oxygen consumption because the other limb remains in a resting position; this is better tolerated by COPD patients experiencing severe dyspnea or fatigue The primary objective of our study is to determine the effectiveness of single-limb resistance exercises in patients with COPD during the exacerbation phase. This research aims to evaluate the potential of this exercise modality to improve the physiological and psychological status of patients during an acute episode.

H0: Single-limb exercise training applied to COPD patients during exacerbation does not change functional exercise capacity compared to the control group.

H1: Single-limb exercise training applied to COPD patients during exacerbation changes functional exercise capacity compared to the control group.

Hypothesis 2:

H02: Single-limb exercise training applied to COPD patients during exacerbation does not change the perception of dyspnea and fatigue compared to the control group.

H2: Single-limb exercise training applied to COPD patients during exacerbation changes the perception of dyspnea and fatigue compared to the control group.

Hypothesis 3:

H03: Single-limb exercise training applied to COPD patients during exacerbation does not change peripheral muscle strength compared to the control group.

H3: Single-limb exercise training applied to COPD patients during exacerbation changes peripheral muscle strength compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

Hospital admission due to an acute COPD exacerbation.

Not currently enrolled in an active pulmonary rehabilitation program.

Absence of any additional neurological disorders.

Exclusion Criteria:

Heart failure classified as New York Heart Association (NYHA) Class III or IV. Unstable mental status (indicated by a Mini-Mental State Examination (MMSE) score of 24).

History of major surgery within the last three months. Presence of malignancies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-09-25 (Estimated)

PRIMARY OUTCOMES:
1. Functional Exercise Capacity | Up to 8 weeks
  30-Second Sit-to-Stand Test (30-sec STS): Functional capacity will be assessed using a chair with a height of 43.2 cm and back support. Patients, with arms crossed over their chests, will be instructed to complete as many full stands as possible within 30 seconds. Two practice trials will be performed before recording the final count.
Dyspnea | Up to 8 weeks
  Modified Medical Research Council (mMRC) Scale: Dyspnea perception during daily activities will be recorded. The five levels of the scale will be explained in detail to the participants to determine their perceived respiratory distress
Muscle Strength Assessment | Up to 8 weeks
  Muscle strength will be measured using a digital dynamometer (Commander Echo Manual Muscle Tester, Lafayette Instrument Co., USA). The best of three consecutive measurements will be recorded

SECONDARY OUTCOMES:
Respiratory Muscle Strength | Up to 8 weeks
  Maximal Inspiratory Pressure (MIP) and Maximal Expiratory Pressure (MEP) will be assessed using a portable manometer (Pony FX, Cosmed, Italy). For MIP, patients will perform a maximal inspiration from residual volume; for MEP, a maximal expiration from total lung capacity. The best of three measurements with less than 10% variability will be recorded
Pulmonary Function Test (PFT) | Up to 8 weeks
  Pulmonary functions will be measured in a seated position using a spirometer. Parameters including FVC (Liter (L)), FEV₁ (Liter (L)), TLC (Liter (L)), PEF (L/s) will be recorded as absolute values and percentages of predicted values based on age, height, weight, and gender
Anxiety and Depression | Up to 8 weeks
  Hospital Anxiety and Depression Scale (HADS): This 14-item scale consists of two subscales (7 items each for anxiety and depression). The Turkish validity and reliability of the scale have been established, and permission for use has been secured
Functional Exercise Capacity | Up to 8 weeks
  6-Minute Walk Test (6MWT): Prior to the test, resting heart rate, blood pressure, oxygen saturation ($SpO_2$), and respiratory rate will be measured. Patients will walk the maximum possible distance on a 30-meter flat indoor course for 6 minutes. Dyspnea and fatigue during the test will be evaluated using the Borg Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Alper Kemal Gürbüz, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No